CLINICAL TRIAL: NCT07137910
Title: An Open-label, Multicenter Phase II Clinical Trial to Evaluate the Efficacy and Safety of AHB-137 Injection in Participants With Chronic Hepatitis B Previously Treated With Nucleos (t) Ide Analogues (NA)
Brief Title: A Study to Evaluate the Efficacy and Safety of AHB-137 Injection in Participants With Chronic Hepatitis B (CHB)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ausper Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB-10-8009
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relevant drug treatment group (Experimental)
  Interventions: Drug: AHB-137
- No relevant drug treatment group (Experimental)
  Interventions: Drug: AHB-137

INTERVENTIONS:
Drug: AHB-137 — AHB-137 will be injected

SUMMARY:
This study is an open-label, multicenter phase II clinical study to evaluate the efficacy and safety of AHB-137 injection in participants with CHB previously treated with NA.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the study and sign the informed consent form;
* 18-65 years of age (including boundary values) ;
* Body mass index met the requirements;
* Participants with CHB who are HBsAg or HBV DNA positive for at least 6 months;
* Meet the relevant requirements for prior medications;
* HBsAg and HBV DNA and liver function indicators meet the requirements;
* Effective contraception as required;

Exclusion Criteria:

* Uncontrolled and stable clinically significant abnormalities other than a history of CHB infection;
* Associated liver disease;
* Any serious infection other than CHB infection requires intravenous anti-infective therapy;
* HCV RNA positive, HIV antibody positive, syphilis positive;
* Abnormal laboratory results;
* Diseases associated with vascular inflammatory conditions;
* QT interval corrected heart rate (Fridericia method) abnormal;
* History of malignancy or ongoing assessment of possible malignancy;
* History of allergies, or allergic constitution;
* Participants with recent major trauma or major surgery, or planning surgery;
* Those who are participating in another clinical trial, or have not undergone a protocol-specified washout period prior to this study;
* Prior/current use of prohibited medications;
* Inappropriate for participation in this trial as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-27 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with persistent HBsAg < limit of detection (LOD) and HBV DNA < lower limit of quantification (LLOQ) at the 24th week after all treatment for CHB was discontinued. | At the 24th week after all treatment for CHB was discontinued

SECONDARY OUTCOMES:
Proportion of participants with persistent HBV DNA < LLOQ . | During the 24-week period after discontinuation of all CHB treatment
Proportion of participants with persistent HBsAg < limit of detection (LOD) and HBV DNA < lower limit of quantification (LLOQ). | Up to 60 weeks
Detection of the concentration of HBsAg, HBsAb, HBV DNA, HBV RNA, HBcrAg, HBeAb,and HBeAg. | Up to 60 weeks
Relapse rate and time after discontinuation of NAs therapy. | Up to 60 weeks
Changes of the score of Health-Related Quality of Life (HBQOL) in participants compared with baseline. | Up to 60 weeks
Changes of the score of EuroQol Five-Dimension Five-Level Scale (EQ-5D-5L) in participants compared with baseline. | Up to 60 weeks
Number and percentage of participants with detectable anti-drug antibodies (ADA). | Up to 60 weeks
Sequencing of the Viral DNA and/or viral RNA analysis for detection of drug resistance in the target region of AHB-137. | Up to 60 weeks
Safety: Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAE) and clinically significant examination results. | Up to 60 weeks
  Examination including laboratory examination, electrocardiogram (ECG) examination.
Plasma concentrations of AHB-137. | Up to 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Principal Investigator — The First Hospital of Jilin University; Yanhua Ding, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- AusperBio Investigational Site, Jilin, Changchun, China

IPD SHARING:
Plan to Share IPD: No